CLINICAL TRIAL: NCT00965432
Title: A Single-Dose, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study in Healthy, Normal Volunteers to Assess the Safety, Tolerability and Pharmacokinetics of STX107
Brief Title: A Single-Dose Study in Normal Volunteers to Assess the Safety, Tolerability and Pharmacokinetics of STX107
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Randall Carpenter, President and CEO, Seaside Therapeutics, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22006
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: STX107
- STX107 (Active Comparator)
  Interventions: Drug: STX107

INTERVENTIONS:
Drug: STX107 — Single dose of an oral suspension

SUMMARY:
The objectives of this study are to determine the safety and tolerability of single oral doses of STX107 and to determine basic pharmacokinetic (PK) parameters following single oral doses of STX107 when administered via an oral suspension

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy males 18-50 years old, inclusive.
* Able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | During the course of the study and for 14 days after completing the study

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States